CLINICAL TRIAL: NCT04039464
Title: Kids MoD PAH Trial: Mono- vs. Duo-Therapy for Pediatric Pulmonary Arterial Hypertension
Brief Title: Mono vs. Dual Therapy for Pediatric Pulmonary Arterial Hypertension
Acronym: MoD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00300590; UG3HL151458 (NIH); UH3HL151458 (NIH); 1U24TR001609 (NIH); 1U24TR004440 (NIH)
Record Dates: First submitted 2019-07-01; First posted 2019-07-31 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Pulmonary Hypertension
MeSH Terms: interventions — Sildenafil Citrate; Bosentan

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monotherapy with Sildenafil Group (Active Comparator): mono-therapy: first-line monotherapy (sildenafil alone) - in pediatric subjects with PAH.
  Interventions: Drug: Mono-Therapy with Sildenafil
- Duo Therapy with Sildenafil + Bosentan Group (Active Comparator): duo-therapy: compare two treatment strategies - first-line combination therapy (sildenafil and bosentan)
  Interventions: Drug: Duo-Therapy with Sildenafil + Bosentan

INTERVENTIONS:
Drug: Mono-Therapy with Sildenafil — The subjects will be randomized to receive sildenafil alone and will undergo study procedures as outlined in section 1.3. There will not be a placebo group.
  Other Names: Revatio monotherapy
  Arms: Monotherapy with Sildenafil Group
Drug: Duo-Therapy with Sildenafil + Bosentan — The subjects will be randomized to receive combination up-front therapy sildenafil and bosentan and will undergo study procedures as outlined in section 1.3. There will not be a placebo group.
  Other Names: Dual therapy with Revatio and Tracleer
  Arms: Duo Therapy with Sildenafil + Bosentan Group

SUMMARY:
The investigators' central hypothesis is that early combination therapy with two PAH-specific oral therapies that have been shown to be well tolerated in the pediatric population, sildenafil and bosentan, will result in better World Health Organization (WHO) functional class at 12 months after initiation of PAH treatment than therapy with sildenafil alone.

DETAILED DESCRIPTION:
A Phase III, randomized, open label, pragmatic trial to compare the safety and efficacy of first-line combination therapy (sildenafil and bosentan) to first-line monotherapy (sildenafil alone) in pediatric subjects with WHO Functional Classes II or III and precapillary pulmonary hypertension of Group 1 (PAH caused by idiopathic, heritable, drugs or toxins, congenital heart disease, or connective tissue disease) or Group 3 (PAH caused by lung disease or hypoxemia) according to the WHO (Nice) classification system. Precapillary pulmonary hypertension will be defined by standard criteria as mean pulmonary artery pressure over 25 mmHg and/or pulmonary vascular resistance index (PVRI) > 3, as well as pulmonary capillary wedge pressure (or left ventricular end diastolic pressure) ≤ 15 mmHg as determined by cardiac catheterization.

For infants less than one year of age for whom cardiac catheterization is not considered as part of the clinical team's recommended approach, enrollment will be possible without catheterization if the following four criteria (i-iv) are met:

i. Two separate echocardiograms clearly demonstrate pulmonary hypertension by at least three of the following metrics

1. Elevated MPA pressure (early diastolic PR peak gradient >20 mmHg)
2. Right ventricular hypertrophy (qualitative as mild to severe)
3. Right atrial enlargement (scales for age will be provided)
4. Elevated right ventricular systolic pressure (>35mmHg) on at least two at least two reliable spectral Doppler envelopes during the echocardiogram and in the setting of normal for age documented systolic blood pressure at least two reliable spectral Doppler envelopes during the echocardiogram
5. Flattening or (R to L) bowing of the interventricular septum (qualitative or by elevated eccentricity index)
6. Diminished RV function (RV fractional area change <35%) and/or TAPSE below published normal range for age and weight;

ii. There is no clinical or imaging evidence of left heart dysfunction;

iii. Pulmonary venous stenosis and atresia are ruled out by CT angiography or MRI unless all four pulmonary veins are unequivocally normal on the two separate echocardiograms;

iv. There is no evidence of hemodynamically significant left-to-right shunting across an unrestricted systemic to pulmonary shunt.

Study subjects will be followed with current standard of care assessments and diagnostics, including longitudinal clinical evaluations, determinations of functional class (FC), serial NT-pro-Brain Natriuretic Peptide (NT-proBNP) levels, and echocardiography. Data from these studies will be analyzed in central core facilities that will be used by all participating study sites.

Clinical endpoints are the focus of this study. However, additional data collection is planned for exploratory aims to examine the potential role for future application of novel metrics of outcomes in children with PAH (e.g., pediatric QOL and actigraphy), as described below. The investigators also plan to collect blood, swab and urine samples to determine whether inherent genomic variations or novel proteomic biomarkers will associate with clinical responsiveness to interventions within the cohort. Bio-specimens will be obtained to further test the hypothesis that therapeutic responders will have a different genomic or proteomic profile as compared to subjects who do not respond well to therapy.

Bio-specimens will include the following:

1. Blood for DNA, peripheral blood mononuclear cells, plasma, and serum; and
2. Paired Box Gene (PAXgene) tubes for RNA and miRNA studies; and
3. Urine for biomarker analysis.

Because sildenafil and bosentan have different mechanisms of action targeting different intracellular pathways, combination therapy is a rational treatment strategy for pediatric patients with PAH. Past work in adult PAH suggests that combination therapy with longer duration agents with the same mechanisms of action may cause greater and more sustained improvement in clinical course in comparison with monotherapy. Whether children with PAH respond and tolerate combination therapy better than monotherapy has not been studied. In addition, despite a growing experience with sequential therapy, additional medications are added only after clinical deterioration or failure to sustain responsiveness.

Pharmacokinetics will be assessed during this study in order to determine whether drug levels or compliance with therapy affect outcomes in this cohort. In addition, pharmacokinetics data and related clinical responses from mono- and dual therapy participants will be compared. Interactions between these agents are well known, whereby bosentan decreases sildenafil levels. As a result, sildenafil levels during mono- and combination therapy will be further defined by the planned pharmacokinetics in the current protocol. In addition to strengthening this current study design, such data will form a basis for optimizing the use of these agents and potential strategies for dose adjustments in the broader scope of clinical care in the future.

ELIGIBILITY:
Inclusion Criteria

* Children who have not been treated with long-term targeted PAH drug therapy, which include calcium channel blockers (CCB); prostanoids, endothelin receptor antagonists (ERA) or PDE-5 inhibitors (PDE5i) (note that agents used for vasoreactivity testing during cardiac catheterization, or for acute periprocedural stabilization will be discontinued prior to study enrollment these include inhaled nitric oxide and/or prostacyclin analogs) a. Children who have been receiving subtherapeutic dosing of sildenafil (and no other standing therapy) for less than 2 weeks at the time of their referral for evaluation at a PH Center, may be included after a washout period of two days. Subtherapeutic is defined as dosage less than those shown in Section 6.1.2 sildenafil dosing chart. If, prior to the initial diagnostic cardiac catheterization, the independent clinical practitioner is planning to stop low dose sildenafil that is judged to not have therapeutic impact on hemodynamics by echocardiography, one may include this candidate for enrollment. These children will be followed closely during the washout period for clinical findings of cardiorespiratory changes, and with echocardiography and NT-proBNP measurements. Abnormal findings on these screening tests will prompt consideration of acute initiation of inhaled nitric oxide therapy. Therapy for pulmonary hypertension as determined by randomization for the study, may be started immediately after the two day washout period.
* Diagnosis of PAH by cardiology diagnostics

  1. Diagnosis by cardiac catheterization with in the previous six months: PAH is defined as the presence of mean pulmonary artery pressure > 25mmHg, pulmonary capillary wedge pressure (or left atrial or left ventricular end diastolic pressure) ≤ 15 mmHg, and pulmonary vascular resistance index (PVRI) > 3 Woods Units
  2. For infants less than one year of age for whom cardiac catheterization is not considered as part of the clinical team's recommended approach, enrollment will be possible without catheterization if the following four criteria are met:

  i. Two separate echocardiograms clearly demonstrate pulmonary hypertension by at least three of the following metrics:
  * Elevated MPA pressure (early diastolic PR peak gradient >20 mmHg)
  * Right ventricular hypertrophy (qualitative as mild to severe)
  * Right atrial enlargement (scales for age will be provided)
  * Elevated right ventricular systolic pressure (>35mmHg) on at least two at least two reliable spectral Doppler envelopes during the echocardiogram and in the setting of normal for age documented systolic blood pressure at least two reliable spectral Doppler envelopes during the echocardiogram.
  * Flattening or (R to L) bowing of the interventricular septum (qualitative or by elevated eccentricity index)
  * Diminished RV function (RV fractional area change <35%) and/or TAPSE below published normal range for age and weight.

ii. There is no clinical or imaging evidence of left heart dysfunction; iii. Pulmonary venous stenosis and atresia are ruled out by CT angiography or MRI unless all four pulmonary veins are unequivocally normal on the two separate echocardiograms; iv. There is no evidence of hemodynamically significant left-to-right shunting across an unrestricted systemic to pulmonary shunt (this is unlikely to be a concern for PFO, small ASD, or restrictive PDA or VSD).

* Age ≥3 months to < 18 years (until just before the 18th birthday);
* WSPH groups 1 or 3 NOT due to unrepaired congenital heart disease (other than a patent foramen ovale), OR single ventricle, OR Eisenmenger's syndrome (PLEASE NOTE that only patients with Group 1.1, 1.2, 1.3, and 1.4.4 or Group 3 PAH will be included and this does not include those with much rarer presentations with connective tissue disease, HIV infection, portal hypertension, schistosomiasis, or persistent PAH of the newborn);
* Current WHO FC II or III.

Exclusion Criteria

* Inability or failure to provide informed consent;
* The presence of syncope, overt RV failure, cyanotic "spells" or systemic hypotension within 4 weeks of enrollment;
* Evidence of diffuse or focal pulmonary venous disease, left-sided heart functional disease;
* Known hypersensitivity to metabolites, or formulation components such as vehicle, preservatives or fillers that are contained in the investigational drugs;
* Pregnancy or breastfeeding;
* Documented history in the medical record of noncompliance with other medical regimens within one year of screening;
* Recent (within 1 year) history of alcohol or illicit drug abuse;
* Participation in any clinical study involving another investigational drug or device within 4 weeks;
* Comorbidities

  a. Disorders treated with cyclosporine A or glyburide

  b. Disorders treated with CYP3A Inhibitors and Beta Blockers

  c. Congenital heart disease that was repaired within 6 months of enrollment;

  i. A repaired patent ductus arteriosus within two months prior to enrollment does not constitute an exclusion.

ii. Anatomic issues with a measured Qp:Qs on cardiac catheterization of 1.3 or less are not considered hemodynamically significant and will therefore not be exclusions (i.e. patent foramen ovale, atrial septal defect, small muscular ventricular septal defect, and patent ductus arteriosus)

* Laboratory values of exclusion at the screening visit

  1. serum ALT or AST lab value that is > 2xULN
  2. serum bilirubin lab value that is > 1.5xULN
  3. creatinine clearance < 30 mL/min;
* Inability to comply with all study procedures and availability for duration of study;
* Inability to take oral medications as prescribed;
* Inability to agree to lifestyle considerations throughout the study (please see section 5.3) and for four weeks thereafter.
* Children over 1 year of age with WSPH group 1 PAH attributed to IPAH or HPAH who are robustly responsive to acute vasodilator testing and who might benefit from a first line trial of oral CCB therapy as assessed by the treating physician and as described in PAH guidelines.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in WHO functional class (FC) of Mono vs. Dual Therapy | Baseline, 12 months
  There are four WHO functional classes: Class I: Pulmonary hypertension without resulting limitation of physical activity; Ordinary physical activity does not cause undue dyspnea or fatigue, or chest pain or near-syncope; Class II: Pulmonary hypertension resulting in a slight limitation of physical activity; Comfortable at rest; Ordinary physical activity causes undue dyspnea or fatigue, or chest pain or near-syncope; Class III: Pulmonary hypertension resulting in a marked limitation of physical activity; Comfortable at rest; Less than ordinary physical activity causes undue dyspnea or fatigue, or chest pain or near-syncope; Class IV: Pulmonary hypertension resulting in inability to carry out any physical activity without symptoms; Signs of right heart failure; Marked limitation of physical activity; Dyspnea and/or fatigue may be present at rest; Discomfort.
  This will be an assessment of a change from one class to another per participant in each arm.

SECONDARY OUTCOMES:
Time to clinical worsening (TTCW) | 24 months
  TTCW has become increasingly used in multicenter randomized clinical trials of adult pulmonary hypertension (PH) and will be used in this trial to capture time (in days) from study enrollment to clinical worsening. Disease progression will be defined as deterioration in WHO FC and the need for additional therapy for subjects less than 8 years of age. Subjects that are over 8 years old will follow adult criteria for this event - both deterioration in WHO FC and more than a 15% decrease in 6 minute walk distance (MWD) from baseline. TTCW is defined as a composite including disease progression, hospitalization for worsening PH, addition of other prostanoid drug therapies, Potts shunt, lung transplantation or atrial septostomy, and all-cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Romer, MD, Principal Investigator — Johns Hopkins University
Locations (10):
- United States (10):
  - Children's Hospital Colorado, Aurora, Colorado
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Johns Hopkins Medical Institutions, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
This study will be conducted in accordance with the following publication and data sharing policies and regulations:
  National Institutes of Health (NIH) Public Access Policy, which ensures that the public has access to the published results of NIH funded research. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive PubMed Central upon acceptance for publication.
  This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals.
Time Frame: 1 year after study completion
Access Criteria: Written request